CLINICAL TRIAL: NCT01978886
Title: Prevalence of Unknown and Known Diabetes in Patients With Frozen Shoulder
Status: Completed | Type: Observational
Sponsor: Sygehus Lillebaelt (Other)
Collaborators: Amager Hospital (Other)
Responsible Party: Principal Investigator, per hviid gundtoft, MD, Ph.D.-student, Sygehus Lillebaelt
Other Study IDs: Gundtoft-01
Record Dates: First submitted 2013-10-26; First posted 2013-11-08 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus; Frozen Shoulder
Keywords: Diabetes Mellitus; frozen shoulder; adhesive capsulitis
MeSH Terms: conditions — Diabetes Mellitus; Bursitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — whole blood for patients not diagnosed with diabetes.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patient with diabetes: Patients who have been diagnoses with diabetes.
- Patients without diabetes: Patients who have not previous been diagnosed with diabetes.

SUMMARY:
The purpose of the study is to investigate how high the prevalence of diabetes (known and unknown) is among patients with a frozen shoulder. Our hypothesis is that it is around 30-40 %.

Another purpose is to investigate whether patients with diabetes have a worse and more painful frozen shoulder than patients without diabetes, and whether the diabetes have an influence on the prognosis.

DETAILED DESCRIPTION:
Patients who are not diagnosed with diabetes would be ask to give a blood sample to investigate if they have an unknown diabetes.

All patients with frozen shoulder will be asked to fill out a questionnaire (Oxford Shoulder Score) to clarify how bad their frozen shoulder is. All patients will receive the questionnaire 6 and 24 month following the date on inclusion.

ELIGIBILITY:
Inclusion Criteria: All newly referred patients who is being diagnosed with frozen shoulder -

Exclusion Criteria: age below 25 or above 75, pt. who don't read or understand danish, not danish citizen, patients with mental illness, pt. with a abuse of alcohol or substances, pregnancy, pt. who within 4 months have been injected with adrenocortical hormone, arthrosis in the glenohumeral joint, avascular necrosis of caput humeri, rotator cuff lesion.

-

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All newly referred patients to one of the involved hospitals who is diagnosed with frozen shoulder.
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2013-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
prevalence of known and unknown diabetes diabetes | 1 year

SECONDARY OUTCOMES:
diabetes influence on the prognosis of frozen shoulder | 24 months
  how the status of diabetes influence the prognosis of frozen shoulder. The patient will be asked to fill out oxford shoulder score at the time of inclusion and at 6 and 24 months follow-up. The two groups (patients with and without diabetes) will be compared using the oxford shoulder score.

CONTACTS AND LOCATIONS:
Overall Officials: per h gundtoft, md, Principal Investigator — Sygehus Lillebaelt
Locations (3):
- Denmark (3):
  - Amager Hospital, Amager, Copenhagen
  - Sygehus Lillebaelt, Kolding, Kolding
  - Vejle Sygehus, Vejle, Vejle

REFERENCES:
- [Derived] Gundtoft PH, Attrup ML, Kristensen AK, Vobbe JW, Sorensen L, Holmich P. Diabetes mellitus affects the prognosis of frozen shoulder. Dan Med J. 2020 Sep 8;67(10):A02200071. PMID 33046203